CLINICAL TRIAL: NCT06018844
Title: Novel mHealth Physical Activity Intervention for Youth With Type 1 Diabetes Mellitus
Status: Terminated | Type: Observational
Why Stopped: PI decision based on reduced staffing and funds.
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: University of Kansas (Other); Nemours Children's Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00002143
Record Dates: First submitted 2023-08-07; First posted 2023-08-31 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: NUDGE — NUDGE is a brief mHealth text messaging intervention designed to promote activity in adolescents by allowing them to set, monitor, and receive feedback on daily PA goals through text message.

SUMMARY:
The goal of this longitudinal cohort study is to learn about a mHealth intervention in Type 1 Diabetes (T1D)

The main question[s] it aims to answer are:

* Does the intervention increase the amount of text messages between the mHealth software and participants?
* Do the text messages from the Nudge software increase moderate to vigorous physical activity (MVPA) in participants?
* Does the MVPA encouraged by the Nudge software improve the HbA1c levels of participants?

Participants will:

* Receive text messages from the Nudge software
* Report physical activity goals via the text messages to the Nudge software
* Wear both an accelerometer and an actigraph for three weeks (spread out across the beginning, 30 days, and 90 days of participation)
* Complete surveys at the beginning of participation
* Complete daily surveys while wearing the devices
* Complete surveys at the end of participation
* Record physical activity in study surveys

ELIGIBILITY:
Inclusion Criteria:

* Participants 12.00-21.99 years old
* Participants with a physician confirmed T1D diagnosis.
* T1D diagnosis was at least 6 months prior to study enrollment
* Participants are on an intensive insulin regiment (either with an insulin pump or multiple daily injection)
* Participants must be using a continuous glucose monitor (CGM)
* Participants and parents/legally authorized representatives (LARS) of participants less than 18.00 speak/read English.

Exclusion Criteria:

* Participants with evidence of type 2 or monogenic diabetes.
* Participants with a comorbid chronic condition (e.g., renal disease).
* Participants with presence of severe psychiatric disorders.
* Participants with a diagnosis of low vision (vision that cannot be corrected with contact lenses or eyeglasses).
* Participants with limited mobility that would prevent participant from engaging in daily physical activity, self-assessed by participant.

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients 12.00 to 21.99 with Type 1 Diabetes
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2024-07-25 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Clements, MD, Principal Investigator — Children's Mercy
Locations (1):
- Children's Mercy, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dabelea D. The accelerating epidemic of childhood diabetes. Lancet. 2009 Jun 13;373(9680):1999-2000. doi: 10.1016/S0140-6736(09)60874-6. Epub 2009 May 27. No abstract available. PMID 19481250
- [Background] Vehik K, Hamman RF, Lezotte D, Norris JM, Klingensmith G, Bloch C, Rewers M, Dabelea D. Increasing incidence of type 1 diabetes in 0- to 17-year-old Colorado youth. Diabetes Care. 2007 Mar;30(3):503-9. doi: 10.2337/dc06-1837. PMID 17327312
- [Background] Mayer-Davis EJ, Dabelea D, Lawrence JM. Incidence Trends of Type 1 and Type 2 Diabetes among Youths, 2002-2012. N Engl J Med. 2017 Jul 20;377(3):301. doi: 10.1056/NEJMc1706291. No abstract available. PMID 28723318
- [Background] Miller GF, Coffield E, Leroy Z, Wallin R. Prevalence and Costs of Five Chronic Conditions in Children. J Sch Nurs. 2016 Oct;32(5):357-64. doi: 10.1177/1059840516641190. Epub 2016 Apr 4. PMID 27044668
- [Background] American Diabetes Association. 13. Children and Adolescents: Standards of Medical Care in Diabetes-2020. Diabetes Care. 2020 Jan;43(Suppl 1):S163-S182. doi: 10.2337/dc20-S013. PMID 31862756
- [Background] Riddell MC, Gallen IW, Smart CE, Taplin CE, Adolfsson P, Lumb AN, Kowalski A, Rabasa-Lhoret R, McCrimmon RJ, Hume C, Annan F, Fournier PA, Graham C, Bode B, Galassetti P, Jones TW, Millan IS, Heise T, Peters AL, Petz A, Laffel LM. Exercise management in type 1 diabetes: a consensus statement. Lancet Diabetes Endocrinol. 2017 May;5(5):377-390. doi: 10.1016/S2213-8587(17)30014-1. Epub 2017 Jan 24. PMID 28126459
- [Background] Miculis CP, De Campos W, da Silva Boguszweski MC. Correlation between glycemic control and physical activity level in adolescents and children with type 1 diabetes. J Phys Act Health. 2015 Feb;12(2):232-7. doi: 10.1123/jpah.2013-0024. Epub 2014 Feb 5. PMID 24508755
- [Background] Nguyen T, Obeid J, Walker RG, Krause MP, Hawke TJ, McAssey K, Vandermeulen J, Timmons BW. Fitness and physical activity in youth with type 1 diabetes mellitus in good or poor glycemic control. Pediatr Diabetes. 2015 Feb;16(1):48-57. doi: 10.1111/pedi.12117. Epub 2014 Jan 20. PMID 24444038
- [Background] Tully C, Aronow L, Mackey E, Streisand R. Physical Activity in Youth With Type 1 Diabetes: a Review. Curr Diab Rep. 2016 Sep;16(9):85. doi: 10.1007/s11892-016-0779-6. PMID 27475093
- [Background] Cushing CC, Mitchell TB, Bejarano CM, Walters RW, Crick CJ, Noser AE. Bidirectional Associations Between Psychological States and Physical Activity in Adolescents: A mHealth Pilot Study. J Pediatr Psychol. 2017 Jun 1;42(5):559-568. doi: 10.1093/jpepsy/jsw099. PMID 28131985
- [Background] Lenhart, A. (2015). Teens, Social Media, & Technology Overview. Retrieved from http://pewinternet.org/2015/04/09/teens-social-media-technology-2015/
- [Background] Fedele DA, Cushing CC, Fritz A, Amaro CM, Ortega A. Mobile Health Interventions for Improving Health Outcomes in Youth: A Meta-analysis. JAMA Pediatr. 2017 May 1;171(5):461-469. doi: 10.1001/jamapediatrics.2017.0042. PMID 28319239
- [Background] Yang CH, Maher JP, Conroy DE. Implementation of behavior change techniques in mobile applications for physical activity. Am J Prev Med. 2015 Apr;48(4):452-5. doi: 10.1016/j.amepre.2014.10.010. Epub 2015 Jan 6. PMID 25576494
- [Background] Brannon EE, Cushing CC. A systematic review: is there an app for that? Translational science of pediatric behavior change for physical activity and dietary interventions. J Pediatr Psychol. 2015 May;40(4):373-84. doi: 10.1093/jpepsy/jsu108. Epub 2014 Dec 13. PMID 25502745
- [Background] Michie S, Abraham C, Whittington C, McAteer J, Gupta S. Effective techniques in healthy eating and physical activity interventions: a meta-regression. Health Psychol. 2009 Nov;28(6):690-701. doi: 10.1037/a0016136. PMID 19916637
- [Background] Militello LK, Melnyk BM, Hekler E, Small L, Jacobson D. Correlates of Healthy Lifestyle Beliefs and Behaviors in Parents of Overweight or Obese Preschool Children Before and After a Cognitive Behavioral Therapy Intervention With Text Messaging. J Pediatr Health Care. 2016 May-Jun;30(3):252-60. doi: 10.1016/j.pedhc.2015.08.002. Epub 2015 Oct 1. PMID 26429638
- [Background] Cushing CC, Bejarano CM, Ortega A, Sayre N, Fedele DA, Smyth JM. Adaptive mHealth Intervention for Adolescent Physical Activity Promotion. J Pediatr Psychol. 2021 Jun 3;46(5):536-546. doi: 10.1093/jpepsy/jsaa125. PMID 33484137
- [Background] Carver CS, Scheier MF. Control theory: a useful conceptual framework for personality-social, clinical, and health psychology. Psychol Bull. 1982 Jul;92(1):111-35. No abstract available. PMID 7134324
- [Background] Cushing CC, Steele RG. A meta-analytic review of eHealth interventions for pediatric health promoting and maintaining behaviors. J Pediatr Psychol. 2010 Oct;35(9):937-49. doi: 10.1093/jpepsy/jsq023. Epub 2010 Apr 14. PMID 20392790
- [Background] Bergenstal RM, Ahmann AJ, Bailey T, Beck RW, Bissen J, Buckingham B, Deeb L, Dolin RH, Garg SK, Goland R, Hirsch IB, Klonoff DC, Kruger DF, Matfin G, Mazze RS, Olson BA, Parkin C, Peters A, Powers MA, Rodriguez H, Southerland P, Strock ES, Tamborlane W, Wesley DM. Recommendations for standardizing glucose reporting and analysis to optimize clinical decision making in diabetes: the Ambulatory Glucose Profile (AGP). Diabetes Technol Ther. 2013 Mar;15(3):198-211. doi: 10.1089/dia.2013.0051. Epub 2013 Feb 28. PMID 23448694
- [Background] Patton SR, Clements MA, Fridlington A, Cohoon C, Turpin AL, Delurgio SA. Frequency of mealtime insulin bolus as a proxy measure of adherence for children and youths with type 1 diabetes mellitus. Diabetes Technol Ther. 2013 Feb;15(2):124-8. doi: 10.1089/dia.2012.0229. Epub 2013 Jan 14. PMID 23317372
- [Background] Laurent J, Catanzaro SJ, Joiner TE, Rudolph KD, Potter KI, Lambert S, Gathright T. A measure of positive and negative affect for children: scale development and preliminary validation. Psychol Assess. 1999; 11: pp. 326.
- [Background] Terry PC, Lane AM, Lane HJ, Keohane L. Development and validation of a mood measure for adolescents. J Sports Sci. 1999 Nov;17(11):861-72. doi: 10.1080/026404199365425. PMID 10585166
- [Background] Levesque CS, Williams GC, Elliot D, Pickering MA, Bodenhamer B, Finley PJ. Validating the theoretical structure of the Treatment Self-Regulation Questionnaire (TSRQ) across three different health behaviors. Health Educ Res. 2007 Oct;22(5):691-702. doi: 10.1093/her/cyl148. Epub 2006 Nov 30. PMID 17138613
- [Background] Nelson TD, Benson ER, Jensen CD. Negative attitudes toward physical activity: measurement and role in predicting physical activity levels among preadolescents. J Pediatr Psychol. 2010 Jan-Feb;35(1):89-98. doi: 10.1093/jpepsy/jsp040. Epub 2009 May 15. PMID 19447878
- [Background] Fox KR, Corbin CB. The physical self-perception profile: development and preliminary validation. J Sport Exerc Psychol. 1989; 11:408-430.
- [Background] Duncan TE, McAuley E. Social support and efficacy cognitions in exercise adherence: a latent growth curve analysis. J Behav Med. 1993 Apr;16(2):199-218. doi: 10.1007/BF00844893. PMID 8315646
- [Background] Motl RW, Dishman RK, Trost SG, Saunders RP, Dowda M, Felton G, Ward DS, Pate RR. Factorial validity and invariance of questionnaires measuring social-cognitive determinants of physical activity among adolescent girls. Prev Med. 2000 Nov;31(5):584-94. doi: 10.1006/pmed.2000.0735. PMID 11071840
- [Background] Lowe MR, Butryn ML, Didie ER, Annunziato RA, Thomas JG, Crerand CE, Ochner CN, Coletta MC, Bellace D, Wallaert M, Halford J. The Power of Food Scale. A new measure of the psychological influence of the food environment. Appetite. 2009 Aug;53(1):114-8. doi: 10.1016/j.appet.2009.05.016. Epub 2009 Jun 12. PMID 19500623
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686

RESULTS

PARTICIPANT FLOW:
Groups:
- Primary Arm: Main group of patients 13.00 to 21.99 with T1D
Period: Overall Study
Arm/Group | Primary Arm
Started | 1
Completed | 0
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Primary Arm
Number analyzed (Participants) | 1
Age, Continuous [Mean (Full Range); unit: years] | 17 [17 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: %Daily Text Messages Exchanged Between Youth and the NUDGE Bot
Description: percent of daily text messages exchanged between youth and the NUDGE bot
Time Frame: Through study completion, an average of 3.5 months
Population: Study terminated before analysis took place, due to slow enrollment and unexpected termination the little data collected could not be analyzed.
Arm/Group | Primary Arm
Number analyzed (Participants) | 0

2. Primary Outcome: Moderate to Vigorous Physical Activity (MVPA) Levels
Description: Participants' MVPA levels
Time Frame: Day 1, 30 and 90
Population: as for outcome 1
Arm/Group | Primary Arm
Number analyzed (Participants) | 0

3. Secondary Outcome: %Days That Youth Wear the Actigraph
Description: Percent of days that youth wear the actigraph
Time Frame: Day 1, 30 and 90
Population: as for outcome 1
Arm/Group | Primary Arm
Number analyzed (Participants) | 0

4. Secondary Outcome: %Daily Physical Activity (PA) Schedules That Participants Complete
Description: percent of daily PA schedules that participants complete
Time Frame: Day 1, 30 and 90
Population: as for outcome 1
Arm/Group | Primary Arm
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in Participant HbA1c
Description: Change in participant HbA1c
Time Frame: Through study completion, an average of 3.5 months
Population: as for outcome 1
Arm/Group | Primary Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 11 months
Arm/Group | Primary Arm
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT06018844/Prot_SAP_000.pdf
  • Informed Consent Form (2024-07-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT06018844/ICF_001.pdf